CLINICAL TRIAL: NCT07359430
Title: An Exploratory, Multi-centre, Two-part Study to Describe Chronic Induced Urticaria Characteristics and Explore Novelbiomarkers With a Multimodal Patient Profiling Approach by Comparing CIndU Patients to Chronic Spontaneousurticaria Patients and Healthy Volunteers
Brief Title: Deep Phenotyping of CIndU
Status: Recruiting | Type: Observational
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: UMC Utrecht (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CHDR2324
Record Dates: First submitted 2025-06-11; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Skin Diseases; Angio-Oedema and/or Urticaria
Keywords: Chronic inducible urticaria; Symptomatic dermographism
MeSH Terms: conditions — Skin Diseases; Chronic Inducible Urticaria; Familial dermographism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples
  * Skin punch biopsies
  * Tape strips of skin surface
  * Swab of skin surface
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Omalizumab: In this treatment arm, a total of 30 patients-comprising 10 with chronic spontaneous urticaria (CSU), 10 with symptomatic dermographism (SD), and 10 with cold urticaria (ColdU)-will receive omalizumab at a dose of 300 mg every 4 weeks.
- Healthy volunteers: As a control group, 10 healthy volunteers without a history of inflammatory skin disease or atopic conditions will be included.

SUMMARY:
Chronic inducible urticaria (CIndU) is a group of skin disorders defined by recurrent itchy or burning wheals or angioedema that recur for more than six weeks with a specific triggering factor. This is different from chronic spontaneous urticaria which does not have a specific triggering factor. CIndU is subclassified in nine subtypes with each having its own specific trigger. These subtypes are further divided in physical urticarias (symptomatic dermographism, cold urticaria, delayed pressure urticaria, solar urticaria, heat urticaria, vibratory angioedema) or non-physical urticarias, i.e., cholinergic urticaria, aquagenic urticaria, and contact urticaria.

Symptomatic dermographism (SD) is the most prevalent subtype of the physical urticarias. Its prevalence in Western populations is estimated to be between 1-5%. Following SD, cold urticaria (ColdU) is the next most common form, its annual incidence is estimated to be 0.05%. In this study, patients with the ColdU and symptomatic SD subtypes will be enrolled.

As of yet, disease diagnosis of SD and ColdU is mostly purely clinical (clinical picture + patients' history), as there is a lack of objective biomarkers. Currently only two objective tools are available for the diagnosis of SD and ColdU, which are the FricTest and Temptest (both provocation tests). In addition, there is a lack of objective biomarkers for the prediction of treatment response and for the monitoring of treatment effects, as this is nowadays only monitored by patient reported outcomes.

DETAILED DESCRIPTION:
The objective of this study is to deep phenotype CIndU (subtype SD and ColdU) and detect novel biomarkers for diagnosis andtreatment response as well as establish methodologies for (non-) invasive monitoring of treatment effects in chronic inducible urticaria.

For this purpose, a study with a multi-modal approach will be performed for in-depth characterization of SD and ColdU. The study willconsist of 2 parts: in part A the biology of disease will be investigated, and in part B the response of the biomarkers to real-world treatment with omalizumab will be monitored (part B). The former to characterize objectively measured disease characteristics and mechanisms underlying its development, the latter to monitor response of the disease and its characteristics to standard of care treatment once in four weeks. The study focusses on cellular, molecular, biophysical, imaging and microbiome analyses in comparisonwith chronic spontaneous urticaria (CSU) patients and matched healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Male and female subjects between 18-69 years of age; in general, stable good health as per judgement of the investigator based upon the results of a medical history, physical examination and vital signs.
* No clinically significant skin disease in the research area
* No history of hypertrophic scarring or keloid.
* Willing to give written informed consent and willing and able to comply with the study protocol.
* Negative TempTest and FricTest at screening.
* Participant is willing to refrain from extensively washing (including bathing, swimming, showering and excessive sweating) the skin 12 hours before study visit 1.

Eligible patients:

* Male and female subjects aged ≥18 years
* Diagnosis of SD, ColdU or CSU (moderate to severe according to international guidelines (Zuberbier et al, 2022)) for ≥3 months and symptomatic disease despite treatment with H1 antihistamines (up to fourfold the approved dose).
* Patients currently on an antihistamine (up to fourfold the approved dose) must be on a stable dose for at least 2 weeks prior to day 1 and must maintain the same stable dose throughout the treatment period. Patients are according to the stepped care model eligible to start treatment with omalizumab
* Willing to give written informed consent and willing and able to comply with the study protocol.
* Positive provocation test:

  1. For ColdU patients: developing a wheal at the test site within 10 min after using TempTest® at any temperature at both screening and Baseline. Alternatively, patients with a negative TempTest® may also be included if they have a positive ice cube test;
  2. For SD patients: developing a wheal at the test site within 10 min after using FricTest® with ≥ 3mm at both screening and Baseline.
* For CSU patients: negative TempTest® and FricTest® at screening
* Participant is willing to refrain from extensively washing (including bathing, swimming, showering and excessive sweating) the skin 12 hours prior to Day 1 and EOS.
* Female participants of reproductive potential must agree to use contraception from screening until EOS.

Exclusion Criteria:

* Significant, uncontrolled or unstable disease in any organ system as per judgment of the investigator (regardless of association with the immunosuppressing disorder/therapy), including but not limited to: psychiatric, neurologic, cardiovascular, pulmonary, gastrointestinal, hepatic, renal, endocrine, hematologic or respiratory disease.
* History of immunological abnormality (e.g., immune suppression) that may interfere with study objectives, in the opinion of the investigator.
* Loss or donation of blood over 500 mL within three months prior to screening.
* Positive hepatitis B surface antigen (HbsAg), hepatitis C antibody (HCV ab), or human immunodeficiency virus antibody (HIB ab) at screening
* Known infection requiring (topical or oral) antibiotic therapy within 56 days prior to Day 1.
* The use of systemic antibiotic therapy for >2 months the past 12 months.
* The use of any oral/systemic medication (e.g. immunomodulatory, immunosuppressive) within 28 days prior to Day 1, if the investigator judges that it may interfere with the study objectives.
* Treatment with omalizumab within 5 half lives (120 days) prior to Day 1
* Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding.
* Have any current and/or recurrent clinically significant or subject reported skin condition other than the CInDU/CSU wherefore subject is included in the study.
* Evidence of current drug or alcohol abuse.
* History of regular alcohol consumption within 12 months of the trial defined as an average weekly intake of >21 alcoholic drinks/week for men or >14 alcoholic drinks/week for women (i.e., 1 drink is equivalent to 150 mL of wine or 360 mL of beer or 45 mL of hard liquor)

Healthy volunteers

- Participation in an investigational drug study within 3 months prior to screening or more than 4 times a year.

Eligible patients

* For CIndU patients: active CSU or other forms of CIndU besides ColdU or SD that may interfere with study assessments. For CSU patients: presence of active CIndU disease that may interfere with study assessments.
* Urticarial or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to C1 inhibitor deficiency).
* Active, pruritic skin condition in addition to CIndU (CIndU patients) or CSU (CSU patients).
* Routine doses of the following medications within 30 days prior to Day 1: Systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide.
* Intravenous (IV) immunoglobulin G (IVIG), or plasmapheresis within 30 days prior to screening.
* Regular (daily/every other day) doxepin (oral) use within 6 weeks prior to Day 1.
* Any H2 antihistamine use within 7 days prior to Day 1.
* Any leukotriene receptor antagonist (LTRA) (montelukast or zafirlukast) within 7 days prior to Day 1.
* Patients with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved.
* Hypersensitivity to omalizumab or any component of the formulation.
* History of anaphylactic shock.
* Evidence of parasitic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Absolute eosiniphil count | Baseline - day 99
  cells/µL
IgG-anti-FcεRI | Baseline - day 99
  IU/mL
Absolute basophil count | Baseline - day 99
  cells/µL
C-reactive protein | baseline - day 99
  mg/L
D-dimer | Baseline - day 99
  µg/mL
Complement assessment | Baseline - day 99
  mg/dL
Total serum IgE | Baseline - day 99
  IU/mL
Basophil activcation test (BAT) | Baseline - day 99
  % activation or Stimulation index
Cytokine profile assessment | Baseline - day 99
  pg/mL
Tissue mass cytometry (CyTOF) | Baseline - day 99
  Skin punch biopsies (4mm) will be taken from (non-)lesional skin and healthy for tissue mass cytometry (CyTOF).
RNA-sequencing analysis | Baseline - day 99
  Skin punch biopsies (4mm) will be taken from (non-)lesional skin and healthy for RNA-sequencing analysis
Next-generation sequencing of skin swabs | Baseline - day 99
  The microbiome is collected by swabbing. The abundance of bacteria is thereafter determined using next-generation sequencing.
Composition and diversity of faecal microbiota | Baseline - day 99
  Faecal samples will be collected to measure the composition and diversity of gut microbiota.
3D Multispectral imaging | Baseline - day 99
  The redness and superficial morphology of (non-)lesional skin sites and healthy skin will be determined using a 3D multispectral imaging system.
Laser Speckle Contrast Imaging (LSCI) | Baseline - day 99
  The cutaneous microcirculation of (non-)lesional skin sites and healthy skin will be monitored over a 40 second timespan with a laser speckle contrast imager.
2D photography | Baseline - day 99
  Standardized 2D clinical photographs will be taken of lesional and non-lesional skin, as well as healthy control skin, to build a longitudinal photo library for visual assessment of disease morphology and treatment response over time.

SECONDARY OUTCOMES:
Urticaria Activity Score over 7 days (UAS7) | Baseline - day 99
  The Urticaria Activity Score over 7 days (UAS7) is a validated patient-reported outcome measure used to assess the severity and frequency of urticaria symptoms-specifically wheals (hives) and pruritus (itch)-over the previous week. Scores range from 0 to 42, with higher scores reflecting more severe disease activity. The UAS7 is applied exclusively in patients with chronic spontaneous urticaria (CSU) to monitor disease burden and evaluate treatment response.
Urticaria Control Test (UCT) | Baseline - day 99
  The Urticaria Control Test (UCT) is a validated patient-reported outcome measure used to assess disease control in patients with chronic spontaneous urticaria (CSU). The total UCT score ranges from 0 to 16, with higher scores indicating better disease control. This questionnaire is used exclusively in patients with CSU to monitor treatment response and disease management over time.
Dermatology Life Quality Index (DLQI) | Baseline - day 99
  The Dermatology Life Quality Index (DLQI) is a validated patient-reported outcome measure that assesses the impact of skin diseases on patients' quality of life over the previous week. The total DLQI score ranges from 0 to 30, with higher scores indicating greater impairment in quality of life. A score of 0 reflects no impact, whereas 30 represents the most severe impact on quality of life. The DLQI will be assessed in all patients across the included skin disease cohorts.
Symptomatic Dermographism Activity Score (SDAS) | Baseline - day 99
  The Symptomatic Dermographism Activity Score (SDAS) is a patient-reported outcome measure specifically designed to assess disease activity in individuals with symptomatic dermographism. Patients rate the severity of their symptoms, such as itching and whealing, over the previous 24 hours on a scale from 0 to 4, with higher scores indicating more severe symptoms. The SDAS will be assessed daily in patients with symptomatic dermographism throughout the study to monitor disease activity and treatment response.
Symptomatic Dermographism Quality of Life Questionnaire (SD-QoL) | Baseline - day 99
  The Symptomatic Dermographism Quality of Life Questionnaire (SD-QoL) is a disease-specific, patient-reported outcome measure that evaluates the impact of symptomatic dermographism on patients' daily functioning and well-being. It covers domains such as symptoms, emotional burden, and social limitations, with higher scores indicating greater impairment in quality of life. The SD-QoL will be administered to all patients with symptomatic dermographism to assess the condition's impact over time and in response to treatment.
Cold Urticaria Activity Score (ColdUAS) | Baseline - day 99
  The Cold Urticaria Activity Score (ColdUAS) is a patient-reported outcome measure used to assess daily disease activity in individuals with cold urticaria. Patients rate the severity of their symptoms, such as itching, whealing, and swelling, over the previous 24 hours on a scale from 0 to 3 for each symptom, with higher scores reflecting greater disease activity. The ColdUAS will be completed daily by patients with cold urticaria throughout the study to monitor fluctuations in disease activity and evaluate treatment effects.
Cold Urticaria Quality of Life Questionnaire (ColdU-QoL) | Baseline - day 99
  The Cold Urticaria Quality of Life Questionnaire (ColdU-QoL) is a disease-specific, patient-reported outcome measure that assesses the impact of cold urticaria on various aspects of daily life, including symptoms, emotional well-being, and social and occupational functioning. Higher scores indicate greater impairment in quality of life. The ColdU-QoL will be administered to all patients with cold urticaria to evaluate the burden of disease and changes in quality of life over the course of treatment.
Activity Tracking Sleep | Baseline - day 99
  Subjects are requested to wear a smartwatch at all times which register sleep (hrs, minutes, seconds of rest)
Activity Tracking Steps | Baseline - day 99
  Subjects are requested to wear a smartwatch at all times which register steps (amount of steps taken)

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Centre for Human Drug Research, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided